CLINICAL TRIAL: NCT04576195
Title: Immediate Neurophysiological Effects of Ultrasound-Guided Percutaneous Electrical Stimulation on Radial Nerve in Patients With Lateral Epicondylalgia
Brief Title: Immediate Neurophysiological Effects of PENS on Radial Nerve in Patients With Lateral Epicondylalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19/043 (b)
Record Dates: First submitted 2020-09-28; First posted 2020-10-06 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-01

CONDITIONS: Tennis Elbow
Keywords: Lateral Epicondylalgia; Lateral Epicondylitis; Lateral Elbow Tendinopathy; Lateral Elbow Pain; Percutaneous Electrical Nerve Stimulation
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real PENS (Experimental): One single session of PENS
  Interventions: Other: Real PENS
- Sham PENS (Sham Comparator): One single session of Sham-PENS
  Interventions: Other: Sham PENS

INTERVENTIONS:
Other: Real PENS — The technique will be performed ultrasound-guided on the radial nerve, the places of the needle's insertions will be the following:
  Needle will be placed at under the lateral intermuscular septum between the triceps brachii and brachialis, approximately 10cm superior to the lateral epicondyle Needle will be placed at the upper third of the forearm on the posterior interosseous nerve after passing the arcade of Frohse's
  The percutaneous electrical stimulation will be realized with a transcutaneous electric nerve stimulation (TENS) current:
  TENS Frequency 2 Hz TENS Pulse width - 250 microseconds Duration - 30 minutes. TENS Intensity - Increased at an intensity of visible motor response of the innervated musculature and maximal tolerable intensity.
  Administration - One single session.
  Arms: Real PENS
Other: Sham PENS — The technique will be performed ultrasound-guided on the radial nerve, the places of the needle's insertions will be the following:
  Needle will be placed at under the lateral intermuscular septum between the triceps brachii and brachialis, approximately 10cm superior to the lateral epicondyle Needle will be placed at the upper third of the forearm on the posterior interosseous nerve after passing the arcade of Frohse's
  The electrical current will not be working, and the needles will be placed during 30 minutes:
  - Administration - One single session
  Arms: Sham PENS

SUMMARY:
Lateral epicondylalgia is a common musculoskeletal condition that approximately affects 1-3% of the general population. Several authors have found greater mechanical pain sensitivity in the radial nerve when compared with healthy subjects. Radial tunnel syndrome exhibits a similar clinical presentation to lateral epicondylalgia. Percutaneous electrical stimulation has shown reduce pain in several conditions. Percutaneous electrical stimulation on the radial nerve could cause an important relief in lateral epicondylalgia.

Hypothesis: Percutaneous electrical stimulation on radial nerve plus in patients with lateral epicondylalgia is better than sham percutaneous electrical stimulation

DETAILED DESCRIPTION:
Randomized, double-blind, placebo controlled clinical trial, using Percutaneous Electrical Nerve Stimulation (PENS). PENS is technique to provide a transcutaneous electrical nerve stimulation current throughout needling filaments place close to the nerve.

Study Aims:

Aim #1: The primary aim of the study is to compare the immediate effect of a single session of PENS on pressure pain sensitivity as measured by pressure pain threshold in patients with lateral epicondylalgia with random assignment to two treatments: PENS or Sham PENS

Aim #2: The secondary aim of the study is to compare the immediate effect on pain free grip strength, on intensity of pain as measured by visual analogue scale (VAS) in patients with lateral epicondylalgia with random assignment to two treatments: PENS or Sham PENS.

ELIGIBILITY:
Inclusion Criteria:

* Lateral epicondylalgia symptoms confirmed with at least 2 of the 4 following test:

  1. pain during palpation of lateral epicondyle
  2. pain on resisted wrist extension
  3. pain on resisted middle finger extension
  4. pain during hand-grip

Exclusion Criteria:

* History of fractures, luxations, surgery and/or musculoskeletal disorders in upper limb.
* Neurological disorders, inflammatory and/or degenerative diseases.
* Having received as treatment techniques that involve needles on the previous 6 months to study enrollment, or having received percutaneous electrical stimulation as a treatment before.
* Cervical pathology, fibromyalgia, unstable cardiovascular diseases, pregnant women or under suspect of pregnancy.
* Contraindications of needle's insertions: anticoagulant therapy, needle phobia, diabetes, hypothyroidism, lymphoedema, muscular diseases).
* Contraindications of electrical current application

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Changes in Pressure pain threshold using an algometer | Baseline and immediate (10 minutes after intervention)
  Measurement of pressure pain threshold in the lateral epicondyle, radial nerve in the spiral groove, C5-C6 zygapophyseal joints, and the tibialis anterior muscle.

SECONDARY OUTCOMES:
Changes in Pain Intensity: Visual Analogue Scale | Baseline and immediate (10 minutes after intervention)
  Pain intensity measured with a 100 mm (0 - No pain - 100 The worst pain) visual analogue scale
Changes in Pain-Free Grip Strength | Baseline and immediate (10 minutes after intervention)
  Measurement the amount of force that the patient generates to the onset of pain as measured with a dynamometer
Changes in Self-perceived Improvement between baseline and follow-up periods | Time Frame: Baseline,10 minutes post-intervention
  Global ratings on changes in regards to their level of elbow well-being since the treatment on a 15-point self-report scale (from -7, very much worse, to 7, completely recover)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Complutense de Madrid, Madrid, Spain